CLINICAL TRIAL: NCT02156830
Title: Multidisciplinary Approach and Counseling of the Obese Patient Before and After Bariatric Surgery: Qualitative Interviews
Brief Title: Multidisciplinary Approach and Counseling of the Obese Patient Before and After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Ina Gesquiere, PhD Student, KU Leuven
Other Study IDs: INOGMA2
Record Dates: First submitted 2013-08-19; First posted 2014-06-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The project consists of qualitative interviews with all the members of the obesity team (endocrinologist, bariatric surgeon, dietician, psychologist,..) in different Flemish hospitals. These interviews have the aim to gain insight into the current practice about counseling patients with bariatric surgery, with a focus on medication counseling. This will make it possible to assess the strengths and weaknesses in the current practice of obese patients who will undergo and have undergone bariatric surgery.

DETAILED DESCRIPTION:
The project consists of qualitative interviews with all the members of the obesity team (endocrinologist, bariatric surgeon, dietician, psychologist,..) in different Flemish hospitals. These interviews have the aim to gain insight into the current practice about counseling patients with bariatric surgery, with a focus on medication counseling. We will do a benchmarking and also qualitative analyses of the interviews using Nvivo 10.

This will make it possible to assess the strengths and weaknesses in the current practice of obese patients who will undergo and have undergone bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* All the members of the obesity team should be prepared to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The different health care professionals of the obesity team
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Difference between multidisciplinary approach in bariatric surgery population in Flanders and the guidelines | The interviews will be performed once
  We will do a benchmarking and a qualitative research to give an overview of the counseling of obese patients before and after bariatric surgery and to identify the barriers of to a multidisciplinary approach in the counseling of bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Foulon, PhD PharmD, Principal Investigator — KU Leuven
Locations (1):
- Ina Gesquiere, Leuven, Belgium